CLINICAL TRIAL: NCT02340767
Title: Decision Aids for the Management of Suspicious Occlusal Caries Lesions
Acronym: SOCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Dental Practice-Based Research Network (Network)
Collaborators: Kaiser Permanente (Other); HealthPartners Institute (Other); The University of Texas Health Science Center at San Antonio (Other); University of Alabama at Birmingham (Other); University of Florida (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-003-E
Record Dates: First submitted 2014-12-30; First posted 2015-01-19 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries
Keywords: Suspicious Occlusal Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No Device Clinicians (No Intervention): The clinicians will not receive any additional training.
- Spectra Device Clinicians (Experimental): The clinicians in the Spectra Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of clinicians familiarizing themselves with the device through unsupervised clinical use with patients.
  Interventions: Device: Spectra Device
- DIAGNOdent Device Practitioners (Experimental): The clinicians in the DIAGNOdent Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of clinicians familiarizing themselves with the device through unsupervised clinical use with patients.
  Interventions: Device: DIAGNOdent

INTERVENTIONS:
Device: Spectra Device — Spectra Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
  Arms: Spectra Device Clinicians
Device: DIAGNOdent — DIAGNOdent Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
  Arms: DIAGNOdent Device Practitioners

SUMMARY:
The study will determine whether clinicians who use a diagnostic device treat suspicious occlusal carious lesions (SOCL) surgically more often, with the same frequency, or less frequently, than dentists not relying on a diagnostic device. The study will also determine -- among those SOCLs that are opened -- whether the proportion of lesions that extend into the dentin when dentists are using a diagnostic device is more than, the same, or less than when no device is used.

DETAILED DESCRIPTION:
The overall objectives of this study is to assess the contributions of diagnostic devices in clinicians' decision-making processes surrounding suspicious occlusal carious lesions (SOCL), an assessment that has not yet been attempted, despite the growing popularity of these devices. SOCLs can be defined as occlusal surface areas where visual, tactile, and radiographic signs are insufficient to definitively diagnose caries but where some of these signs are present.This study examines the use of two diagnostic devices on dental practitioners' identification and treatment of SOCLs.

During a four-week pre-intervention period, 90 clinicians will collect and record descriptive and treatment information for the SOCLs they identify. Clinicians will then be randomized into one of 3 study arms: no diagnostic device, DIAGNOdent®, and Spectra®, and will collect and record similar information as the pre-intervention period for another six weeks, enrolling an additional 20 SOCLs. They will also complete diagnostic vignettes at the beginning and end of the study, as well as a post-study questionnaire on the utility of the devices, if assigned to a device arm. Analyses will examine differences in proportion of SOCLs treated surgically in the groups with and without the diagnostic device; and, for those treated surgically, differences in the proportions of SOCLs with extension into dentin. Differences in pre- and post-study responses on the vignettes will suggest which components of the decision-making process involved in SOCL identification and management have been modified by use of the diagnostic devices.

ELIGIBILITY:
Inclusion Criteria:

Practitioner: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Is enrolled in the National Dental Practice Based Research Network (National Dental PBRN);
* Has completed an Enrollment Questionnaire;
* Is a general or pediatric dentist who is licensed in the United States to treat patients and treats patients in the United States on a recurring basis;
* Is trained and certified in Human Subjects Protection Training;
* Has attended or viewed a National Dental PBRN orientation session or attended at least one annual regional meeting of practitioners or has attended a National Dental PBRN workshop at the International Association for Dental Research (IADR) or American Association for Dental Research (AADR).
* Performs restorative dentistry routinely in their practices as reported on the enrollment questionnaire;
* Has no clinical experience (no history of routine use in practice within the past one year) with either of the devices being used in the study and declares no conflict of interest with the corporations that produce DIAGNOdent® and Spectra®; and
* Is able to complete the pre-and post-study vignettes online.

Practice: If a practitioner is in a practice where they share an operatory (including a hygiene chair) only 1 dentist can be recruited from that practice.

Patient: In order to be eligible to participate in this study, an individual with a SOCL must meet all of the following criteria:

* Willing to provide consent according to regionally approved procedures and/or obtain parent/legal guardian permission as applicable;
* Willing to comply with all study procedures; Is six years of age or older; and
* Has not participated in the study previously. Patients will be enrolled only once throughout the study (this includes the pre-intervention and intervention phases for the pilot study and full study).

Tooth: In order to be eligible to be included in this study, a tooth with a SOCL must meet all of the following criteria:

* Permanent tooth;
* No radiographic evidence of caries into dentin based on available radiographs;
* Caries into dentin is suspected due to roughness, surface opacities, or staining;
* No symptoms of sensitivity to sweets, cold, air, etc.;
* No restoration on the occlusal surface; and
* No sealant on occlusal surface.

Exclusion Criteria:

* Under the age of 6 years old
* Primary Teeth
* Evidence of Caries into dentin based on available radiographs
* Sensitivity to sweets, cold, air etc.;
* Restoration on the occlusal surface
* Sealant on occlusal surface

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3085 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Study Director — University of Alabama at Birmingham; Sonia K Makhija, DDS, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - HealthPartners Institute for Education and Research, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Dental Practice-Based Research Network — http://NationalDentalPBRN.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had a pre-intervention phase, 108 clinicians (HS trained, consented, and met eligibility criterion) and 1500 patients enrolled. 85 clinicians met the enrollment threshold and were randomized.1500 patients were in the post-intervention phase.The pre- and post patients were not the same so the number analyzed for each group varies.
Groups:
- No Device Practitioners: The practitioners will not receive any additional training.
- Spectra Device Practitioners: The practitioners in the Spectra Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
  Spectra Device: Spectra Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
- DIAGNOdent Device Practitioners: The practitioners in the DIAGNOdent Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
  DIAGNOdent: DIAGNOdent Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
- Pre-intervention Patients no Device; Pre-randomization Patients Spectra; Pre-randomization Patients DIANGOdent; Post-randomization Patients no Device; Post-randomization Patients Spectra; Post-randomization Patients DIAGNOdent: The patients in the pre-intervention group were not the same as the one in the post-intervention group. The clinicians were the same.
Period: Overall Study
Arm/Group | No Device Practitioners | Spectra Device Practitioners | DIAGNOdent Device Practitioners | Pre-intervention Patients no Device | Pre-randomization Patients Spectra | Pre-randomization Patients DIANGOdent | Post-randomization Patients no Device | Post-randomization Patients Spectra | Post-randomization Patients DIAGNOdent
Started | 28 | 28 | 29 | 500 | 474 | 526 | 525 | 444 | 531
Completed | 28 | 28 | 29 | 500 | 474 | 526 | 525 | 444 | 531
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These were the patients in each arm for the pre-intervention and post-intervention. The pre-intervention patients were placed in their group that the clinician was ultimately randomized to. Clinicians were the same pre and post.
Groups:
- No Device Patients Pre-intervention; Spectra Device Patients Pre-intervention; DIAGNOdent Device Patients Pre-intervention: All pre-and post-intervention patients were different, which is why the numbers don't match. We place the pre-intervention patients into the arm their clinican was ultimately assigned to.
- No Device Clinicians: They received no device at randomization
- Spectra Clinicians: The practitioners in the Spectra Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
- DIAGNOdent Clinicians: The practitioners in the DIAGNOdent Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
- Total: Total of all reporting groups
Arm/Group | No Device Patients Pre-intervention | Spectra Device Patients Pre-intervention | DIAGNOdent Device Patients Pre-intervention | No Device Clinicians | Spectra Clinicians | DIAGNOdent Clinicians | No Device Patients Post-intervention | Spectra Device Patients Post-intervention | DIAGNOdent Device Patients Post-intervention | Total
Number analyzed (Participants) | 500 | 474 | 526 | 28 | 28 | 29 | 525 | 444 | 531 | 3085
Age, Continuous [Mean (Standard Deviation); unit: years] — The pre-intervention phase had 1500 patients and the post-intervention had 1500 patients. The pre-intervention patients are not the same as the patients in post-intervention. The clinicians were the same in both phases. Age was not reported for clinicians, only year of graduation. The race collected on the clinician was different as well. I have reported on the information we have collected.
  years
    All patients and clinicians | 32.3 (17.5) | 30.1 (17.0) | 34.7 (17.3) | NA (NA) — This information was not collected on the clinicians, only patients | NA (NA) — This information was not collected on the clinicians, only patients | NA (NA) — This information was not collected on the clinicians, only patients | 37.2 (19.2) | 36.3 (16.1) | 34.7 (16.8) | 36.0 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The pre-intervention patients were different than the post-intervention patients. Clinicians were the same.
  Participants
    All patients and clinicians: Female | 303 | 252 | 328 | 11 | 10 | 12 | 297 | 269 | 302 | 1784
    All patients and clinicians: Male | 197 | 222 | 198 | 17 | 18 | 17 | 228 | 175 | 229 | 1301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patients at the pre-intervention stage are not the same patients as post-randomization, which is why the numbers are different in both phases. Clinicians were the same.
  Participants
    Patients and Clinicians: Hispanic or Latino | 77 | 73 | 84 | 0 | 0 | 1 | 60 | 20 | 51 | 366
    Patients and Clinicians: Not Hispanic or Latino | 395 | 391 | 417 | 26 | 26 | 28 | 443 | 400 | 450 | 2576
    Patients and Clinicians: Unknown or Not Reported | 28 | 10 | 25 | 2 | 2 | 0 | 22 | 24 | 30 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The patients at pre-intervention are not the same patients at post-intervention. We just placed them in the eventual categories. The clinicians were the same.
  Participants
    Patients and Clinicians: American Indian or Alaska Native | 6 | 4 | 9 | 1 | 0 | 0 | 14 | 15 | 17 | 66
    Patients and Clinicians: Asian | 16 | 21 | 21 | 3 | 4 | 6 | 7 | 1 | 2 | 81
    Patients and Clinicians: Native Hawaiian or Other Pacific Islander | 0 | 4 | 2 | NA — This information was not collected on the clinicians, only patients | NA — This information was not collected on the clinicians, only patients | NA — This information was not collected on the clinicians, only patients | 4 | 2 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients and Clinicians: Black or African American | 85 | 72 | 76 | 2 | 1 | 3 | 55 | 66 | 85 | 445
    Patients and Clinicians: White | 353 | 322 | 378 | 21 | 20 | 18 | 407 | 348 | 388 | 2255
    Patients and Clinicians: More than one race | 11 | 11 | 6 | NA — This information was not collected on the clinicians, only patients | NA — This information was not collected on the clinicians, only patients | NA — This information was not collected on the clinicians, only patients | 9 | 4 | 7 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patients and Clinicians: Unknown or Not Reported | 29 | 40 | 34 | 1 | 3 | 2 | 29 | 8 | 31 | 177
Region of Enrollment [Number; unit: patients and clinicians]
  United States | 500 | 474 | 526 | 28 | 28 | 29 | 525 | 444 | 531 | 3085
Number of Patients and Clinicians [Count of Participants; unit: Participants] | 500 | 474 | 526 | 28 | 28 | 29 | 525 | 444 | 531 | 3085

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions That Received Invasive Treatment and the Number of Lesions Receiving Invasive Treatment That Extended Into Dentin
Description: There was one lesion/patient.
Time Frame: Pre-intervention and post-intervention (one day visit)
Population: Only the patients who received invasive treatment were analyzed for extension into dentin.Not all columns add up to the total N due to missing values.
Measure: Number; unit: lesions
Groups:
- No Device Patients in Pre-intervention: The patients in pre-intervention are different than post-intervention.
- No Device Patients Post-intervention; Spectra Patients Post-intervention; DIAGNOdent Patients Post-intervention: The patients in the pre-intervention stage are not the same as the post-intervention stage.
Arm/Group | No Device Patients in Pre-intervention | No Device Patients Post-intervention | Spectra Patients Post-intervention | DIAGNOdent Patients Post-intervention
Number analyzed (Participants) | 1500 | 525 | 444 | 531
lesions
  Invasive (yes/no) : Yes | 603 | 246 | 213 | 248
  Invasive (yes/no) : No | 885 | 277 | 226 | 276
  Extended into dentin : Yes: number analyzed (Participants) | 566 | 227 | 207 | 221
  Extended into dentin : Yes | 349 | 151 | 133 | 144
  Extended into dentin : No: number analyzed (Participants) | 566 | 525 | 444 | 531
  Extended into dentin : No | 217 | 76 | 74 | 77

2. Secondary Outcome: Number of Clinicians in Likelihood of Surgically Treating Lesions in Online Vignettes That Display Two Levels of Five Cues (Color, Surface Smoothness, Surface Luster, Caries Risk, and Device Reading (if Applicable) in Post-intervention
Description: Clinicians' likelihood of treating surgical lesions depicted with brown verses black, smooth verses rough, shiny verses matte, in patients with high verses low caries risk, by post-intervention phases. The outcome measure will be to see what cues were used or treatment decisions in the post-intervention phase. Please note that more than one cue could be chosen, so values may add up to more than 100 percent. Participants in the no device group did not receive a device reading cue.
Time Frame: Post-intervention (dentists completed the vignettes one time)
Measure: Count of Participants; unit: Participants
Arm/Group | No Device Practitioners | Spectra Device Practitioners | DIAGNOdent Device Practitioners
Number analyzed (Participants) | 28 | 28 | 29
Participants
  Luster | 15 | 14 | 12
  Color | 15 | 12 | 11
  Risk | 13 | 10 | 18
  Feel of the lesion | 11 | 10 | 10
  Device reading | 0 | 23 | 27

3. Secondary Outcome: Number of Clinicians in Likelihood of Surgically Treating Lesions in Online Vignettes That Display Two Levels of Four Cues (Color, Surface Smoothness, Surface Luster, and Caries Risk) in Pre-intervention
Description: Clinicians' likelihood of treating surgical lesions depicted with brown verses black, smooth verses rough, shiny verses matte, in patients with high verses low caries risk, by post-intervention phases. The outcome measure will be to see what cues were used or treatment decisions in the pre-intervention phase. Please note that more than one cue could be chosen, so values may add to more than 100 percent of participants.
Time Frame: Pre-intervention (dentists completed the vignettes one time)
Population: Pre-intervention the dentists were not randomized and had no device training and all dentists were combined
Measure: Count of Participants; unit: Participants
Arm/Group | No Device Practitioners
Number analyzed (Participants) | 85
Participants
  Luster | 49
  Color | 40
  Risk | 29
  Feel of the lesion | 31

ADVERSE EVENTS:
Groups:
- No Device Clinicians: The practitioners will not receive any additional training.
- Spectra Device Clinicians: The practitioners in the Spectra Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
  Spectra Device: Spectra Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
- DIAGNOdent Device Clinicians: The practitioners in the DIAGNOdent Device Arm will be trained to the device according to the manufacturers' usual care for training. The training will consist of viewing the manufacturer's instructions for the device. Training will also consist of practitioners familiarizing themselves with the device through unsupervised clinical use with patients.
  DIAGNOdent: DIAGNOdent Caries detection device is used for study data collection recording the results of the dental examination and recording results of dental treatment.
- No Device Patients (Pre-intervention and Post-intervention): The total number of patients in these two phases is 1000 and 0/1000 were affected. These were 2 different sets of patients.
- Spectra Patients (Pre-intervention and Post-intervention): The total number of patients in these two phases is 918 and 0/918 were affected. These were 2 different sets of patients.
- DIAGNOdent Patients (Pre-intervention and Post-intervention): The total number of patients in these two phases is 1057 and 0/1057 were affected. These were 2 different sets of patients.
Arm/Group | No Device Clinicians | Spectra Device Clinicians | DIAGNOdent Device Clinicians | No Device Patients (Pre-intervention and Post-intervention) | Spectra Patients (Pre-intervention and Post-intervention) | DIAGNOdent Patients (Pre-intervention and Post-intervention)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/29 | 0/1000 | 0/918 | 0/1057
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/29 | 0/1000 | 0/918 | 0/1057
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/29 | 0/1000 | 0/918 | 0/1057

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No